CLINICAL TRIAL: NCT05728281
Title: Recommended Time to Resume Sexual Activity After Hysterectomy: Impact on Sexual Function (FSFI® Score) and Complication Rate ISHYS Study
Brief Title: Impact of Time on Sexual Function (FSFI® Score) After Hysterectomy
Acronym: ISHYS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Angers (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 2022-A02714-39
Record Dates: First submitted 2023-02-04; First posted 2023-02-15 (Actual); Last update posted 2025-07-23 (Actual); Status verified 2025-07

CONDITIONS: Time Between Hysterectomy and Resumption of Sexual Relations; Sexual Function
Keywords: benign gynaecological disease; hysterectomy; sexual function; FSFI® score

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Resumption of sexual intercourse recommended 4 weeks after hysterectomy (Other)
  Interventions: Other: Recommended time after hysterectomy
- Resumption of sexual intercourse recommended 8 weeks after hysterectomy (Other)
  Interventions: Other: Recommended time after hysterectomy

INTERVENTIONS:
Other: Recommended time after hysterectomy — Currently there is no consensus on the optimal time to resume sexual activity. Using a randomization, we will therefore compare two groups: one, whose postoperative instructions will indicate a resumption of sexual activity from 4 weeks after the operation and the other from 8 weeks postoperatively. The primary endpoint is the FSFI® score. The patients will answer the FSFI® questionnaire preoperatively and then at 3 months after surgery.

SUMMARY:
In France, more than 62 000 hysterectomies are performed each year. Female sexual function is the result of multiple psychological, social and physiological factors. There is no information in the current literature about the optimum time between the surgery and the sexual relation resumption. The primary outcome is to assess the impact of advising time between hysterectomy and sexual relation resumption by using FSFI® score. Secondaries outcomes are: to describe and compare post-operative complications in the two groups of the study, to describe the follow-up of the recommendation concerning time between surgery and sexual relation resumption and to describe why this recommendation was not followed. This study is based on 4 questionnaires: FSFI® pre-operative and post-operative, pre-operative questionnaire and post-operative questionnaire. This is a monocentric, comparative, of superiority, randomised and prospective study. Patients are randomised into two groups: sexual relation resumption advised 4 weeks after surgery, or 8 weeks. The inclusion criteria are more than 18 years, francophone, in sexual activity, scheduled for a total hysterectomy for benign indication (menometrorrhagia, fibroma, adenomyosis, endometriosis, pelvic floor disorders, low-grade endometrial cancer), considering vaginal, laparoscopic and abdominal approach, and a written consent. Non-inclusion criteria are illiteracy, cognitive disorders, without social security, deprived liberty by judicial or administrative decision, psychiatric care, patient with legal protection, patient incapable of giving consent. If our conclusions confirmed our hypothesis, it can improve clinical practices by providing additional informations for surgeon and patient, to undergo this surgery as serenely as possible.

ELIGIBILITY:
Inclusion Criteria:

* Patient ≥ 18 years old,
* Francophone,
* Sexually active,
* Receiving a conservative or non-conservative total hysterectomy for benign pathology*,
* Having signed a consent form. All surgical approaches are considered, laparoscopic approach with laparoscopic or vaginal closure, vaginal approach and laparotomy.

  *The indications for the procedure selected for this study include:
* Menometrorrhagia,
* Fibroids,
* Adenomyosis,
* Endometriosis,
* Pelvic statics disorder,
* Cervical dysplasia,
* Endometrial cancer not requiring lymph node dissection or additional treatment.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 142 (Estimated)
Dates: Start 2023-06-05 (Actual); Primary Completion 2026-06-05 (Estimated); Study Completion 2026-10-05 (Estimated)

PRIMARY OUTCOMES:
The Female Sexual Function Index score | one year
  Assessment of the impact of the recommended time between hysterectomy and resumption of sexual intercourse on sexual function using the Female Sexual Function Index score

SECONDARY OUTCOMES:
Postoperative complications | one year
  Describe and compare postoperative complications according to the recommended time between hysterectomy and resumption of sexual intercourse. The postoperative complications studied include dyspareunia, spontaneous pain outside of sexual intercourse, metrorrhagia, infection, and vaginal fundal suture release.
Follow-up to the recommendation | one year
  Describe the follow-up to the recommendation in terms of time to resume sexual intercourse and describe the reasons for not following the recommendation

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital of Angers, Angers, France